CLINICAL TRIAL: NCT05353101
Title: Efficiency and Safety of Cyclosporine 0.05% Eye Drops for Vernal Keratoconjunctivitis: a Non-randomized Controlled Study
Brief Title: Cyclosporine 0.05% Eye Drops for Vernal Keratoconjunctivitis Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Yifeng Yu, Deputy chief physician of Ophthalmology center of the Second Affiliated Hospital of Nanchang University, Second Affiliated Hospital of Nanchang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2020] No. (080)
Record Dates: First submitted 2022-04-24; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2021-04

CONDITIONS: Vernal Keratoconjunctivitis; Cyclosporine 0.05% Eye Drops
Keywords: Cyclosporine 0.05% eye drops; Vernal Keratoconjunctivitis; Immunomodulator; Olopatadine Hydrochloride Eye Drops
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Cyclosporine; Ophthalmic Solutions; Loteprednol Etabonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cyclosporine 0.05% eye drops group (Experimental): The patients with VKC will receive Cyclosporine 0.05% eye drops or Loteprednol Etabonate 0.5% and Tobramycin Eye Drops 0.3% effect of Cyclosporine 0.05% eye drops would be evaluated during the follow-up visits.
  Interventions: Drug: Cyclosporine 0.05% eye drops; Drug: Loteprednol Etabonate 0.5% and Tobramycin Eye Drops 0.3%

INTERVENTIONS:
Drug: Cyclosporine 0.05% eye drops — Use of 0.05% CSA could significantly reduce IL-4, IL-5, IL-17A, and TNF in tears of VKC patients- α、 IFN- γ And eosinophil chemokine levels. Cyclosporine A (CSA) can effectively control ocular inflammation by blocking Th2 lymphocyte proliferation and IL-2 production. It can also inhibit the recruitment of eosinophils by inhibiting the release of histamine by mast cells and reducing the production of IL-5 further to improve its curative effect on VKC
Drug: Loteprednol Etabonate 0.5% and Tobramycin Eye Drops 0.3% — Corticosteroids can inhibit the release of mast cells, block the chemotaxis of inflammatory cells, and reduce the number of mast cells and eosinophils in the conjunctiva. At the same time, it can inhibit phospholipase A2 and quickly alleviate symptoms and signs.

SUMMARY:
To observe and compare the clinical efficacy of cyclosporine 0.05% eye drops with Loteprednol Etabonate 0.5% and Tobramycin Eye Drops 0.3% in the treatment of Vernal Keratoconjunctivitis in developing regions of China.

DETAILED DESCRIPTION:
Vernal keratoconjunctivitis (VKC) is an allergic disease that severely affects the eyesight of adolescents. Vernal keratoconjunctivitis (VKC) usually occurs in temperate regions such as the Mediterranean region, the Middle East, Africa, Central America, and the Indian subcontinent. In the EU an estimated 3.2 per 10,000 inhabitants (0.03%). It occurs repeatedly and mainly involves type I and type IV hypersensitivity. long-term standardized treatment is necessary. Therefore, this research aims to compare the readily available cyclosporine 0.05% eye drops and Loteprednol Etabonate 0.5% and Tobramycin Eye Drops 0.3% in developing regions of Asia (China, Jiangxi Province) for long-term drug use in VKC patients in developing countries provide evidence.

ELIGIBILITY:
Inclusion criteria

* patients had a noticeable seasonal, and recurrent Itching, Discomfort(burning, stinging, and foreign body sensation), Photophobia and tears, Viscous discharge;
* Slit-lamp microscopy showed Conjunctival Hyperemia, Tarsal papillary, Limbal hypertrophy, Horner-Trantas dots, Keratitis in some patients;
* No other medication history in recent 2 weeks;
* Patients have high compliance and are willing to take drugs on time and return to the clinic in time

Exclusion criteria:

* with other related immune diseases or other drug use history in recent 2 weeks;
* Patients with evident and severe organic diseases or mental diseases;
* Low compliance, unable to take drugs on time or fail to return to the clinic on time.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Changes of ocular signs | Day 0#7#15#30 and 60d
  The eye signs of the patients were observed under a slit lamp, including Conjunctival Hyperemia, Tarsal papillary, Limbal hypertrophy, Horner-Trantas dots, and Keratitis in some patients.The observer gives the corresponding score.The higher the score, the more serious it is (0-4 points)
Changes of self-conscious symptoms | Day 0#7#15#30 and 60d
  The VAS scoring table was used for the patients' self-conscious symptoms, including pruritus, foreign body sensation, Photophobia and tears, and viscous secretions. The patients under study were self-scored at each review. 0-100 points, 0 indicates no discomfort, and 100 indicates the most significant pain. The intraocular pressure at each review was recorded by a non-contact tonometer.

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No